CLINICAL TRIAL: NCT05488223
Title: Effect of Two Omega 3 Polyunsaturated Fatty Acid Schemes on Insulin Resistance and the Inflammatory and Lipid Profile in Obese Children
Brief Title: Supplementation With PUFA´s in Obese Children
Acronym: PUFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Collaborators: Centro Universitario del Sur, Guadalajara (Unknown); Instituto de Servicios Descentralizados de Salud Pública del Estado de Campeche (Unknown)
Responsible Party: Principal Investigator, Jenny Vilchis Gil, Principal Investigator, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HIM/2013/0001
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Child Obesity; Insulin Resistance; Metabolic Complication
Keywords: child; obesity; insulin resistance; metabolic profile; PUFA ω-3
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Obesity | interventions — Fatty Acids, Monounsaturated

STUDY DESIGN:
Intervention Model Description: Subject to written informed consent, children who agreed to participate were randomly assigned to the following treatment groups. Group 1. Two daily capsules of ω-3FAs; Group 2. Two daily capsules, one of ω-3FAs of 0.9 g + 1 capsule of avocado oil (AcAg) of 0.9 g and; Group 3. Two daily capsules of 0.9 g of AcAg.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Preparation of the intervention products, to blind the study. ω-3 PUFAs (Triple Strength Fish Oil®) were purchased in advance, each capsule contained 540 mg of eicosapentaenoic acid (20:5 n-3) and 360 mg of docosahexaenoic acid (22:6 n-3), for a 0.9g total. Likewise, a commercial brand of avocado oil (AcAg) was purchased in advance, putting the same amount in each capsule. The appearance of the ω-3 PUFA capsules and the AcAg capsules were the same. Then we worked with the company that prepared the blinding of the treatments, packaging bottles of 30 capsules each, labeling them as bottles A and B. The design contemplated giving each child two bottles, one marked to take it for breakfast and another marked to take it with food.
  The content of each of the capsules was saved as a code that was unknown to the participants, the care provider, or the researchers. The codes were opened until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PUFA ω-3 (1.8g/day) (Experimental): ω-3 PUFAs (Triple Strength Fish Oil®) were purchased in advance, each capsule contained 540 mg of eicosapentaenoic acid (20:5 n-3) and 360 mg of docosahexaenoic acid (22:6 n-3), for a 0.9g total. Children and parents were told that they should take 2 capsules of ω-3 PUFAs daily, that is, they took 1.8g/day.
  Parents and children were informed that the duration of the study would be 5 months, in the first three months, the children should take the capsules of the assigned treatment; in the fourth and fifth months they should continue their surveillance with the researchers. At the beginning, they were given 2 bottles of 30 capsules each, identified as formula A or B, according to the assigned group, and they were given a calendar sheet indicating that they should cross out a box if they had consumed the breakfast capsule and cross out another box if the consumed during the meal; Likewise, they were asked to write down any adverse effect, if any, on the same sheet.
  Interventions: Dietary Supplement: AGPI ω-3 (Triple Strength Fish Oil®)
- PUFAs ω-3 0.9 g/day + MUFAs (avocado oil) 0.9 g/day. (Active Comparator): A commercial brand of avocado oil (MUFA) was purchased in advance by putting 0.9g in each capsule. The appearance of the ω-3 PUFA capsules and the avocado oil capsules were the same. Then we worked with the company that prepared the blinding of the treatments, packaging bottles of 30 capsules each, labeling them as bottles A and B. The design contemplated giving each child two bottles, one marked to take it for breakfast and another marked to take it with food. The child was instructed to take 1 capsule per day of PUFA ω-3 (0.9g/d) and 1 capsule of avocado oil (0.9g/d)
  Interventions: Dietary Supplement: AGPI ω-3 + MUFA (avocado oil)
- MUFAs (avocado oil) 1.8 g/day. (Placebo Comparator): The child was instructed to take 2 capsules per day, 1.8g of avocado oil per day.
  Interventions: Dietary Supplement: MUFA (avocado oil) (1.8g)

INTERVENTIONS:
Dietary Supplement: AGPI ω-3 (Triple Strength Fish Oil®) — The children met at a clinical studies office every month for the 5 months, in order to exchange the empty bottles for the full ones and review the consumption record sheet and receive their advice on their diet. In case of absence, the children were located to avoid losses. Finally, at each visit, all the children and their parents received counseling to promote the acquisition of healthy habits related to eating and physical activity, but did not indicate caloric restriction diets or undergo exercise programs.
  Arms: PUFA ω-3 (1.8g/day)
Dietary Supplement: AGPI ω-3 + MUFA (avocado oil) — AGPI ω-3 (0.9g) + MUFA (avocado oil) (0.9g) The children met at a clinical studies office every month for the 5 months, in order to exchange the empty bottles for the full ones and review the consumption record sheet and receive their advice on their diet. In case of absence, the children were located to avoid losses. Finally, at each visit, all the children and their parents received counseling to promote the acquisition of healthy habits related to eating and physical activity, but did not indicate caloric restriction diets or undergo exercise programs.
  Arms: PUFAs ω-3 0.9 g/day + MUFAs (avocado oil) 0.9 g/day.
Dietary Supplement: MUFA (avocado oil) (1.8g) — MUFA (avocado oil) (1.8g) The children met at a clinical studies office every month for the 5 months, in order to exchange the empty bottles for the full ones and review the consumption record sheet and receive their advice on their diet. In case of absence, the children were located to avoid losses. Finally, at each visit, all the children and their parents received counseling to promote the acquisition of healthy habits related to eating and physical activity, but did not indicate caloric restriction diets or undergo exercise programs.
  Arms: MUFAs (avocado oil) 1.8 g/day.

SUMMARY:
Introduction. Insulin resistance (IR) accompanies practically half of children with obesity. This alteration is the border between what can be reversible or permanent. Among the comorbidities associated with IR are T2D and cardio and cerebrovascular diseases, which are the leading causes of death in Mexico. It has been said that the prevention of obesity rather than its treatment is the way to contain this problem. It has been proposed to supplement obese children with IR with ω-3 polyunsaturated fatty acids (PUFA) or ω-9 monounsaturated fatty acids (MUFA) to determine their ability to reverse these alterations.

Objetive. To evaluate the effect of supplementing PUFA ω-3, PUFA ω-9 or both, on the change in anthropometric and metabolic parameters in obese children with IR.

Methods. Clinical trial, randomized triple-blind, in which obese children with IR participated. Intervention. Three groups were integrated that received one of the following treatments for three months: Group 1: PUFA ω-3 1.8 g/day; Group 2: PUFA ω-3 0.9 g/day + PUFA ω-9 0.9 g/day (avocado oil). Group 3: MUFA ω-9 1.8 g/day. Tracing. For 2 more months he continued his clinical surveillance. Anthropometric and metabolic profile measurements were made at baseline, 3 and 5 months. Throughout the study, all three child groups received nutritional counseling, but no calorie-restricted diets or exercise programs were used.

DETAILED DESCRIPTION:
Specific objectives

1. To compare between the study groups, the concentrations of glucose, insulin and HOMA-IR Index, at baseline, at the end of supplementation with PUFA ω-3 and PUFA ω-9 (3 months) and 2 months after supplementation. the supplementation.
2. To compare between the study groups, the concentrations of total cholesterol, HDL cholesterol, LDL cholesterol and TG at baseline, at the end of supplementation and 2 months after supplementation.
3. To compare between the study groups the change in the percentile values of body mass index (BMI) and waist circumference (WC), between the study groups, at baseline, at the end of supplementation (3 months) and 2 months after supplementation.

Methods. A randomized, controlled, triple-blind clinical trial was conducted, which included 133 children with obesity (BMI ≥95th percentile) and with IR (HOMA-IR ≥ 3.0).

ELIGIBILITY:
Inclusion Criteria:

* Children with obesity (BMI ≥95 pc), according to the CDC reference tables.
* HOMA-IR ≥ 3.0.
* That they grant their written consent to participate.

Exclusion Criteria:

* Patients with any chronic disease.
* Patients who consume medications that alter their metabolic profile.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Change in insulin resistance | Change in insulin resistance from baseline at 3 months
  Insulin concentrations were immunoassayed with MILLIPLEX® MAP, based on automated Luminex xMAP® technology. Luminex that uses microsphere techniques, which are coated with specific capture antibodies, and employs two fluorescent dyes. The bioassay result was quantified based on the fluorescence signals. The data was integrated and analyzed with the MILLIPLEX® Analyst 5.1 software.
  The following equation was used to obtain the homeostasis model to assess the index of insulin resistance (HOMA-IR): fasting glucose (mg/dl) x fasting insulin (μU/ml) / 405
Change in insulin resistance | Change in insulin resistance from baseline at 5 months
  Insulin concentrations were immunoassayed with MILLIPLEX® MAP, based on automated Luminex xMAP® technology. Luminex that uses microsphere techniques, which are coated with specific capture antibodies, and employs two fluorescent dyes. The bioassay result was quantified based on the fluorescence signals. The data was integrated and analyzed with the MILLIPLEX® Analyst 5.1 software.
  The following equation was used to obtain the homeostasis model to assess the index of insulin resistance (HOMA-IR): fasting glucose (mg/dl) x fasting insulin (μU/ml) / 405
Change in BMI percentile | Change in BMI percentile from baseline at 3 months
  Weight (kg) and height (cm) were taken using internationally accepted procedures and standardized per person. Briefly, weight and height were measured without shoes and in light clothing. Weight was taken with a digital scale (Seca 884, Hamburg, Germany) with a precision of 0.1 kg; height was measured using a stadiometer (Seca 225). With the values of weight, height, age and sex, the BMI percentile was obtained according to the CDC.
Change in BMI percentile | Change in BMI percentile from baseline at 5 months
  Weight (kg) and height (cm) were taken using internationally accepted procedures and standardized per person. Briefly, weight and height were measured without shoes and in light clothing. Weight was taken with a digital scale (Seca 884, Hamburg, Germany) with a precision of 0.1 kg; height was measured using a stadiometer (Seca 225). With the values of weight, height, age and sex, the BMI percentile was obtained according to the CDC.

SECONDARY OUTCOMES:
Change in waist circumference (percentile) | Change in waist circumference percentile from baseline at 3 months
  Waist circumference (cm) was measured with the children in a standing position, using a flexible tape measure (Seca 201®), placed at the midpoint between the lower rib and the iliac crest after a normal exhalation, according to the protocol of WHO. Using the tables of waist circumference of Mexican children, a very high risk was considered if the circumference was greater than the 90th percentile
Change in waist circumference (percentile) | Change in waist circumference percentile from baseline at 5 months
  Waist circumference (cm) was measured with the children in a standing position, using a flexible tape measure (Seca 201®), placed at the midpoint between the lower rib and the iliac crest after a normal exhalation, according to the protocol of WHO. Using the tables of waist circumference of Mexican children, a very high risk was considered if the circumference was greater than the 90th percentile.
Change in metabolic parameters (mg/dL) | Change in metabolic parameters (mg/dL)from baseline at 3 months
  Glucose (mg/dL), low-density lipoprotein (mg/dL), high-density lipoprotein (mg/dL), triglycerides (mg/dL), and total cholesterol (mg/dL) determinations were analyzed with enzymatic methods according to the procedures manual of the Central Laboratory of the Hospital Infantil de México Federico Gómez (Dimension-RXL, Dade Behring, Germany).
Change in metabolic parameters (mg/dL) | Change in metabolic parameters (mg/dL) from baseline at 5 months
  Glucose (mg/dL), low-density lipoprotein (mg/dL), high-density lipoprotein (mg/dL), triglycerides (mg/dL), and total cholesterol (mg/dL) determinations were analyzed with enzymatic methods according to the procedures manual of the Central Laboratory of the Hospital Infantil de México Federico Gómez (Dimension-RXL, Dade Behring, Germany).
Change in cytokines (pg/mL) | Change in cytokines (pg/mL) from baseline at 3 months
  In serum, the following cytokines IL1B, IL4, IL_6, IL10, IFNg, MCP1, TNTa and Leptin (pg/mL) are determined. Based on automated Luminex xMAP® technology.
Change in cytokines (pg/mL) | Change in cytokines (pg/mL) from baseline at 5 months
  In serum, the following cytokines IL1B, IL4, IL_6, IL10, IFNg, MCP1, TNTa and Leptin (pg/mL) are determined. Based on automated Luminex xMAP® technology.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Vilchis Gil, PhD, Principal Investigator — Hospital Infantil de Mexico Federico Gomez
Locations (1):
- Hospital Infantil de México Federico Gómez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared once the statistical analyzes are carried out and it is sent for publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: When the study is published, the database will be available in the journal indefinitely.
Access Criteria: Access to the database through the journal where it is published, in the supplementary files section

REFERENCES:
- [Result] Juarez-Lopez C, Klunder-Klunder M, Madrigal-Azcarate A, Flores-Huerta S. Omega-3 polyunsaturated fatty acids reduce insulin resistance and triglycerides in obese children and adolescents. Pediatr Diabetes. 2013 Aug;14(5):377-83. doi: 10.1111/pedi.12024. Epub 2013 Feb 25. PMID 23438101
- [Result] Juarez-Lopez C, Klunder-Klunder M, Medina-Bravo P, Madrigal-Azcarate A, Mass-Diaz E, Flores-Huerta S. Insulin resistance and its association with the components of the metabolic syndrome among obese children and adolescents. BMC Public Health. 2010 Jun 7;10:318. doi: 10.1186/1471-2458-10-318. PMID 20529295
- [Result] Vilchis-Gil J, Galvan-Portillo M, Klunder-Klunder M, Cruz M, Flores-Huerta S. Food habits, physical activities and sedentary lifestyles of eutrophic and obese school children: a case-control study. BMC Public Health. 2015 Feb 11;15:124. doi: 10.1186/s12889-015-1491-1. PMID 25885348
- See also: This page is from the Hospital Infantil de México Federico Gómez where the research protocol was approved and developed. — http://himfg.com.mx/